CLINICAL TRIAL: NCT07303075
Title: Family-Centred Acceptance and Commitment Therapy After Paediatric Acquired Brain Injury
Brief Title: Family-Centred ACT After Paediatric ABI
Acronym: FamilyCARE-ABI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24080
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Acquired Brain Injury
Keywords: Paediatric; Acceptance and Commitment Therapy; Psychological Flexibility; Acquired Brain Injury; Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): The only arm of the study - dyads will receive treatment (ACT)
  Interventions: Other: Acceptance and Commitment Therapy (DNA-V)

INTERVENTIONS:
Other: Acceptance and Commitment Therapy (DNA-V) — Family-Centred ACT for ABI will begin with a needs assessment and comprise needs- and ABI-specific psychoeducation and ACT principles using the DNA-V model of ACT.

SUMMARY:
Children and young people with acquired brain injury (ABI) commonly experience long-term emotional, behavioural, and participation difficulties that can affect quality of life for both them and their families. Parents and caregivers also often experience high levels of stress and reduced wellbeing. Despite these needs, family-centred psychological interventions remain limited. Acceptance and Commitment Therapy (ACT) is a values-focused cognitive-behavioural approach designed to increase psychological flexibility and has shown promise for children with long-term health conditions and for parents of children with ABI, but it has not been directly evaluated as a joint therapeutic approach for children with ABI and their parents.

This study (Family CARE-ABI) evaluates the feasibility, acceptability, and preliminary effectiveness of delivering ACT simultaneously to a young person aged 11-18 with an ABI and their parent/guardian. Up to six dyads will be recruited. The study uses a non-concurrent, multiple-baseline, single-case experimental design in which dyads are randomised to begin a 12-week ACT intervention after either a 3- or 4-week baseline period. Sessions (up to 12, one hour each) are delivered via Microsoft Teams by a trainee clinical psychologist under specialist supervision. Therapy integrates the DNA-V model of ACT-developed for young people-with ABI-specific psychoeducation and skills practice tailored to each dyad's needs.

Outcome measures include mental health and wellbeing (Outcome Rating Scale), psychological flexibility (CompACT or AFQ-Y8), symptoms of anxiety and depression (GAD-7, PHQ-9, or RCADS-25), community participation (CASP/CASP-Y), and needs after ABI (MANTIC). Measures are collected at baseline, post-intervention, and 12-week follow-up, with weekly wellbeing ratings throughout participation. Therapeutic alliance (SRS) is obtained after each intervention session. All dyads will also take part in separate qualitative interviews exploring their experiences of the intervention and its impact.

Safety is closely monitored, including assessment of distress, adverse events, and any safeguarding concerns. Participation is voluntary, and dyads may withdraw at any time without affecting usual care. Data are stored securely and anonymised for analysis.

The study aims to generate early evidence regarding whether family-centred ACT may support psychological wellbeing, flexibility, and participation for young people with ABI and their parents, and to inform future intervention development and larger-scale trials.

ELIGIBILITY:
Inclusion Criteria Both the CYP-ABI and parent participants must meet the inclusion criteria to be recruited to the study.

CYP-ABI participant inclusion criteria include:

* Aged 11 to 18 years at time of recruitment.
* Living at home with parent/guardian.
* Received treatment for an ABI.
* Have sufficient cognitive ability to engage with therapy sessions.
* Has capacity to provide verbal or written informed consent (aged 16 and above) or assent (aged 15 and younger).
* Has the ability to speak sufficient English to understand and engage with the therapeutic and research materials
* Consents for parent/guardian participant involvement in study.

Parent participant inclusion criteria include:

* Aged > 18 at time of recruitment. There is no upper age limit.
* Has the ability to speak sufficient English to understand and engage with the therapeutic and research materials
* Has capacity to provide verbal or written informed consent for self and CYP participant.

Exclusion Criteria:

CYP-ABI and parent participant exclusion criteria include:

• CYP or parent participants are currently accessing or have accessed structured psychological intervention within 6 months of study recruitment.

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-12-05 (Estimated); Primary Completion 2026-06-27 (Estimated); Study Completion 2026-06-27 (Estimated)

PRIMARY OUTCOMES:
Outcome Rating Scale | From enrollment to the end of the study at 24 weeks
  Measure of wellbeing

SECONDARY OUTCOMES:
CompACT | Baseline (week 1), following therapy (week 15 or 16), at follow-up (week 24)
  Measure of psychological flexibility for adults
Avoidance and Fusion Questionnaire | Baseline (week 1), following therapy (week 15 or 16), at follow-up (week 24)
  Measure of psychological flexibility for children
GAD & PHQ9 | Baseline (week 1), following therapy (week 15 or 16), at follow-up (week 24)
  Measures of adult anxiety and depression
RCADS | Baseline (week 1), following therapy (week 15 or 16), at follow-up (week 24)
  Measure of child anxiety and depression
CASP/CASP-Youth Version | Baseline (week 1), following therapy (week 15 or 16), at follow-up (week 24)
  Measure of child participation
MANTIC | Baseline (week 1), following therapy (week 15 or 16), at follow-up (week 24)
  Measure of needs after acquired brain injury
Session Rating Scale | Baseline (week 1), following therapy (week 15 or 16), at follow-up (week 24)
  Measure of therapeutic alliance

IPD SHARING:
Plan to Share IPD: No